CLINICAL TRIAL: NCT03493386
Title: A Single Centre, Single Dose, Open-label, Randomised, 2-way Crossover Study in Healthy Japanese Male Subjects to Evaluate the Bioequivalence of Daprodustat Tablets (2 mg Tablet vs. 4 mg Tablet) (Part 1) and the Food Effect on the Pharmacokinetics of Daprodustat (Part 2)
Brief Title: Daprodustat Bioequivalence and Food Effect Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 207727
Record Dates: First submitted 2018-04-04; First posted 2018-04-10 (Actual); Results first posted 2019-08-06 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-06

CONDITIONS: Anaemia
Keywords: Japan; Crossover; Daprodustat; Bioequivalence; Pharmacokinetics
MeSH Terms: conditions — Anemia | interventions — GSK1278863; Tablets

STUDY DESIGN:
Intervention Model Description: This study will be conducted in two parts. Part 1 is the bioequivalence part in which subjects will receive single dose of 2 tablets of 2 mg daprodustat and single dose of 1 tablet of 4 mg daprodustat in crossover manner. Part 2 is Food effect part. In this part, subjects will receive single dose of 4 mg daprodustat tablet in fasting and fed state in a crossover manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment Group A: Part 1 (Experimental): Subjects will be randomized to receive single dose of two tablets of 2 mg daprodustat in Period 1 and in Period 2 subjects will receive single dose of 4 mg daprodustat. There will be a wash-out period of 5 days between the Periods.
  Interventions: Drug: Daprodustat 2 mg tablet; Drug: Daprodustat 4 mg tablet
- Treatment Group B: Part 1 (Experimental): Subjects will be randomized to receive single dose of 4 mg daprodustat in Period 1 and in Period 2 subjects will receive single dose of two tablets of 2 mg daprodustat. There will be a wash-out period of 5 days between the Periods.
  Interventions: Drug: Daprodustat 2 mg tablet; Drug: Daprodustat 4 mg tablet
- Treatment Group C: Part 2 (Experimental): Subjects will be randomized to receive single dose of 4 mg daprodustat in fed state during Period 1 and in Period 2 subjects will receive single dose of 4 mg daprodustat in fasted state. There will be a wash-out period of 5 days between the Periods.
  Interventions: Drug: Daprodustat 4 mg tablet
- Treatment Group D: Part 2 (Experimental): Subjects will be randomized to receive single dose of 4 mg daprodustat in fasted state during period 1 and in Period 2 subjects will receive single dose of 4 mg daprodustat in fed state. There will be a wash-out period of 5 days between the Periods.
  Interventions: Drug: Daprodustat 4 mg tablet

INTERVENTIONS:
Drug: Daprodustat 2 mg tablet — Daprodustat is available as 2 mg tablet. Subjects will receive daprodustat orally as tablet. A single dose of 2 tablets of 2 mg daprodustat will be administered in a fasted state during Part 1 of the study.
  Arms: Treatment Group A: Part 1; Treatment Group B: Part 1
Drug: Daprodustat 4 mg tablet — Daprodustat is available as 4 mg tablet. Subjects will receive daprodustat orally as tablet. A single dose of 4 mg daprodustat will be administered in a fasted state during Part 1 and in fed and fasted state in Part 2 of the study.

SUMMARY:
This is two-way crossover study to compare pharmacokinetic (PK) of daprodustat 2 milligram (mg) versus 4 mg tablets and food effect on the PK of daprodustat following single oral doses in healthy Japanese male subjects. This study will be conducted in two parts. Part 1 is the bioequivalence part in which subjects will receive single dose of 2 tablets of 2 mg daprodustat and single dose of 1 tablet of 4 mg daprodustat in crossover manner. Part 2 is Food effect part. In this part, subjects will receive single dose of 4 mg daprodustat tablet in fasting and fed state in a crossover manner. There will 5-day wash-out period between each intervention period. There will be approximately 52 subjects in Part 1 and 12 subjects in Part 2. The study will last for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 20 to 55 years of age inclusive, at the time of signing the informed consent.
* Japanese subjects who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Body weight > = 50 kilogram (kg) and body mass index (BMI) within the range 18.5 - 24.9 kilogram per meter square (kg/m^2).
* Male subjects.
* Subjects capable of giving signed informed consent.

Exclusion Criteria:

* History or presence of cardiovascular(CV), respiratory, hepatic, renal, gastrointestinal (GI), endocrine, haematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* Abnormal blood pressure as determined by the investigator.
* ALT >1.5x upper limit of normal (ULN).
* Bilirubin >1.5xULN
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QTcF > 500 millisecond (msec). The QTcF is the QT interval corrected for heart rate according to Fridericia's formula, machine-read or manually over-read. The specific formula that will be used to determine eligibility and discontinuation for an individual subject should be determined prior to initiation of the study. In other words, several different formulae cannot be used to calculate the QT correction (QTc) for an individual subject and then the lowest QTc value used to include or discontinue the subject from the trial.
* The values of Hgb at screening: >=16.0 gram per deciliter (g/dL).
* History of deep vein thrombosis, pulmonary embolism or other thrombosis related condition.
* History of myocardial infarction (MI) or acute coronary syndrome, stroke or transient ischemic attack.
* Subjects that have undergone cholecystectomy.
* History of malignancy within the prior 2 years or currently receiving treatment for cancer.
* Any evidence of heart failure, as defined by the New York Heart Association (NYHA) functional classification system.
* Past or intended use of over-the-counter or prescription medication including vitamins, diet foods and herbal medications within 14 days prior to first dosing.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Current enrolment or past participation (that is administration of last dose of investigational study intervention) within the last 30 days (or 5 half-lives, whichever is longer) before signing of consent in this clinical study involving an investigational study intervention or any other type of medical research.
* The subject with positive serological test for syphilis (Rapid Plasma Reagin [RPR] and Treponema pallidum haemagglutination test [TPHA]), Human immunodeficiency virus (HIV) Antigen/Antibody, Hepatitis B surface antigen (HBsAg), Hepatitis C virus (HCV) antibody, or Human T-cell lymphotropic virus type 1 (HTLV-1) antibody at screening.
* Positive pre-study drug screen.
* Regular alcohol consumption within 6 months prior to the study defined as:for an average weekly intake of >14 units for males. One unit is equivalent to 350 milliliter (mL) of beer, 150 mL of wine or 45 mL of 80 proof distilled spirits.
* Smoking or history of regular use of tobacco- or nicotine-containing products (example nicotine patch, electronic cigarette) within 6 months prior to screening.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.
* History of donation of blood or blood products >= 400 mL within 3 months or >= 200 mL within 1 month prior to the first dosing day.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Japanese male subjects who will be overtly healthy as determined by medical evaluation will be included in the study.
Enrollment: 64 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2018-06-09 (Actual); Study Completion 2018-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20369

REFERENCES:
- [Background] Yamada M, Osamura M, Ogura H, Onoue T, Wakamatsu A, Numachi Y, Caltabiano S, Mahar KM. A Single-Dose, Open-Label, Randomized, Two-Way Crossover Study in Healthy Japanese Participants to Evaluate the Bioequivalence and the Food Effect on the Pharmacokinetics of Daprodustat. Clin Pharmacol Drug Dev. 2020 Nov;9(8):978-984. doi: 10.1002/cpdd.793. Epub 2020 Apr 6. PMID 32250021

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A single center, single dose, open-label, randomized, 2-way crossover study in healthy Japanese male participants to evaluate the bioequivalence of daprodustat tablets, study was conducted at one center in Japan.
Pre-assignment Details: Total 64 healthy participants were enrolled in the study which was conducted from 24-April-18 to 09-June-18, study was conducted in two parts, Part 1 was the bioequivalence of daprodustat Tablets and part 2 was food effect on the pharmacokinetics (PK) of daprodustat.
Groups:
- Part 1: Daprodustat 2mg*2+ Daprodustat 4mg*1: Participants received a single dose Daprodustat 2 milligram (mg) two tablets followed by Daprodustat 4 mg single tablet, administered orally on Day 1.There was a washout period of at least 5 days between the 2 intervention periods.
- Part 1: Daprodustat 4mg*1 + Daprodustat 2mg*2: Participants received a single dose Daprodustat 4 mg one tablet followed by Daprodustat 2 mg two tablets, administered orally on Day 1. There was a washout period of at least 5 days between the 2 intervention periods.
- Part 2: Daprodustat 4mg*1 (Fed) + Daprodustat 4mg*1 (Fast): Participants received a single dose Daprodustat 4 mg one tablet in fed state followed by Daprodustat 4 mg one tablet as single dose in fasted state, administered orally on Day 1.There was a washout period of at least 5 days between the 2 treatment periods.
- Part 2: Daprodustat 4mg*1 (Fast) + Daprodustat 4mg*1 (Fed): Participants received a single dose Daprodustat 4 mg one tablet in fasted state followed by Daprodustat 4 mg one tablet as single dose in fed state, administered orally on Day 1.There was a washout period of at least 5 days between the 2 treatment periods.
Period: Part 1, Intervention Period 1 (2 Days)
Arm/Group | Part 1: Daprodustat 2mg*2+ Daprodustat 4mg*1 | Part 1: Daprodustat 4mg*1 + Daprodustat 2mg*2 | Part 2: Daprodustat 4mg*1 (Fed) + Daprodustat 4mg*1 (Fast) | Part 2: Daprodustat 4mg*1 (Fast) + Daprodustat 4mg*1 (Fed)
Started | 26 | 26 | 0 | 0
Completed | 26 | 26 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 1, Washout Period (at Least 5 Days)
Arm/Group | Part 1: Daprodustat 2mg*2+ Daprodustat 4mg*1 | Part 1: Daprodustat 4mg*1 + Daprodustat 2mg*2 | Part 2: Daprodustat 4mg*1 (Fed) + Daprodustat 4mg*1 (Fast) | Part 2: Daprodustat 4mg*1 (Fast) + Daprodustat 4mg*1 (Fed)
Started | 26 | 26 | 0 | 0
Completed | 26 | 25 | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Part 1, Intervention Period 2 (2 Days)
Arm/Group | Part 1: Daprodustat 2mg*2+ Daprodustat 4mg*1 | Part 1: Daprodustat 4mg*1 + Daprodustat 2mg*2 | Part 2: Daprodustat 4mg*1 (Fed) + Daprodustat 4mg*1 (Fast) | Part 2: Daprodustat 4mg*1 (Fast) + Daprodustat 4mg*1 (Fed)
Started | 26 | 25 | 0 | 0
Completed | 26 | 25 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 2, Intervention Period 1 (2 Days)
Arm/Group | Part 1: Daprodustat 2mg*2+ Daprodustat 4mg*1 | Part 1: Daprodustat 4mg*1 + Daprodustat 2mg*2 | Part 2: Daprodustat 4mg*1 (Fed) + Daprodustat 4mg*1 (Fast) | Part 2: Daprodustat 4mg*1 (Fast) + Daprodustat 4mg*1 (Fed)
Started | 0 | 0 | 6 | 6
Completed | 0 | 0 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Part 2, Washout Period (at Least 5 Days)
Arm/Group | Part 1: Daprodustat 2mg*2+ Daprodustat 4mg*1 | Part 1: Daprodustat 4mg*1 + Daprodustat 2mg*2 | Part 2: Daprodustat 4mg*1 (Fed) + Daprodustat 4mg*1 (Fast) | Part 2: Daprodustat 4mg*1 (Fast) + Daprodustat 4mg*1 (Fed)
Started | 0 | 0 | 6 | 6
Completed | 0 | 0 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Part 2, Intervention Period 2 (2 Days)
Arm/Group | Part 1: Daprodustat 2mg*2+ Daprodustat 4mg*1 | Part 1: Daprodustat 4mg*1 + Daprodustat 2mg*2 | Part 2: Daprodustat 4mg*1 (Fed) + Daprodustat 4mg*1 (Fast) | Part 2: Daprodustat 4mg*1 (Fast) + Daprodustat 4mg*1 (Fed)
Started | 0 | 0 | 6 | 6
Completed | 0 | 0 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Participants Part 1: Participants received daprodustat 2mg*2 tablets and daprodustat 4mg*1 tablets (fasted state) in either of the two treatment periods separated by a washout of at least 5 days between the two treatment periods.
- Total Participants Part 2: Participants received daprodustat 4mg*1 tablet (fed state) and daprodustat 4mg*1 tablet (fasted state) in either of the two treatment periods separated by a washout of at least 5 days between the two treatment periods.
- Total: Total of all reporting groups
Arm/Group | Total Participants Part 1 | Total Participants Part 2 | Total
Number analyzed (Participants) | 52 | 12 | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.9 (6.91) | 30.0 (7.51) | 28.3 (7.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 52 | 12 | 64
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian -Japanese Heritage | 52 | 12 | 64

OUTCOME MEASURES:

1. Primary Outcome: Part 1:Area Under Plasma Concentration-time Curve (AUC) From Zero Hours to Last Measurable Concentration (AUC[0-t]) and AUC From Zero Hours Extrapolated to Infinity AUC [0-inf] of Daprodustat
Description: Blood samples were collected at indicated timepoints and PK analysis was performed. PK parameters were determined by non-compartmental methods with Phoenix WinNonlin version 6.3. PK population comprised of all participants in the Safety population (all randomized participants) who received at least one dose of study intervention) who had at least 1 non-missing PK assessment.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12 hours post-dose on Day 1, 24 hours post-dose on Day 2
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram/milliliter
Groups:
- Part 1: Daprodustat 2mg*2: Participants received a single dose of daprodustat 2mg*2 tablets, administered orally in fasted state on Day 1 in either of period 1 and Period 2 as per the randomization schedule
- Part 1: Daprodustat 4mg*1: Participants received single dose of Daprodustat 4mg one tablet, administered orally in fasted state on Day 1 in either of Period 1 and Period 2 as per randomization schedule
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
Hour*nanogram/milliliter
  AUC (0-t) | 182.8420 (30.7) | 179.6940 (30.4)
  AUC (0-inf) | 183.0240 (30.7) | 179.8710 (30.4)
Statistical Analysis 1: Comparison: Part 1: Daprodustat 2mg*2 vs Part 1: Daprodustat 4mg*1; Test type: Equivalence — If the 90% CI of the ratio of geometric mean doesn't fall within a range of 0.80 to 1.25 i.e., null hypothesis is not rejected the bioequivalence is established if the point estimate falls within a range of 0.90 to 1.11; Ratio of geometric mean = 1.02, 90% CI 2-sided [0.97 to 1.07] — AUC (0-t)
Statistical Analysis 2: Comparison: Part 1: Daprodustat 2mg*2 vs Part 1: Daprodustat 4mg*1; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric mean = 1.02, 90% CI 2-sided [0.97 to 1.07] — AUC(0-inf)

2. Primary Outcome: Part 1:Maximum Observed Drug Concentration (Cmax) of Daprodustat
Description: Blood samples were collected at indicated timepoints and pharmacokinetic (PK) analysis was performed. PK parameters were determined by non-compartmental methods with Phoenix WinNonlin version 6.3.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12 hours post-dose on Day 1, 24 hours post-dose on Day 2
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
Nanogram/milliliter | 88.8811 (37.0) | 85.1365 (37.0)
Statistical Analysis 1: Comparison: Part 1: Daprodustat 2mg*2 vs Part 1: Daprodustat 4mg*1; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric mean = 1.04, 90% CI 2-sided [0.97 to 1.12] — Cmax

3. Primary Outcome: Part 1:Terminal Phase Half-life (T1/2) of Daprodustat and Mean Residence Time (MRT)
Description: Blood samples were collected at indicated timepoints and PK analysis was performed. PK parameters were determined by non-compartmental methods with Phoenix WinNonlin version 6.3.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12 hours post-dose on Day 1, 24 hours post-dose on Day 2
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
hour
  t1/2 | 3.2427 (14.9) | 3.2579 (11.8)
  MRT | 2.8142 (25.9) | 2.9637 (23.2)

4. Primary Outcome: Part 1: Time of Occurrence of Cmax (Tmax) of Daprodustat
Description: as for outcome 3
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12 hours post-dose on Day 1, 24 hours post-dose on Day 2
Population: PK Population
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
hour | 2.000 [1.00 to 4.00] | 2.000 [1.00 to 4.00]

5. Primary Outcome: Part 1: Percentage of AUC (0-inf) Obtained by Extrapolation (Percentage AUCex)
Description: as for outcome 3
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12 hours post-dose on Day 1, 24 hours post-dose on Day 2
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUCex
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
Percentage of AUCex | 0.0862 (53.5) | 0.0836 (55.3)

6. Primary Outcome: Part 1:Apparent Clearance (CL/F) of Daprodustat
Description: as for outcome 3
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12 hours post-dose on Day 1, 24 hours post-dose on Day 2
Population: Safety Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
Liters per hour | 21.8551 (30.7) | 22.2382 (30.4)

7. Primary Outcome: Part 1:Apparent Oral Volume of Distribution (Vz/F) of Daprodustat
Description: as for outcome 3
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12 hours post-dose on Day 1, 24 hours post-dose on Day 2
Population: Safety Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliters (mL)
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
Milliliters (mL) | 102244.3 (33.2) | 104522.8 (30.8)

8. Primary Outcome: Part 1: Elimination Rate Constant (Kel) of Daprodustat
Description: as for outcome 3
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12hours post-dose on Day 1, 24hours post-dose on Day 2
Population: Safety Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per hour
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
Per hour | 0.2138 (14.9) | 0.2128 (11.8)

9. Primary Outcome: Part 2:AUC[0-t] andAUC [0-inf] of Daprodustat
Description: as for outcome 3
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12hours post-dose on Day 1, 24hours post-dose on Day 2
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram/milliliter
Groups:
- Daprodustat 4mg (Fed): Participants received a single dose of daprodustat 4mg one tablet, administered orally in fed state on Day 1 in intervention period 1
- Daprodustat 4mg(Fasted): Participants received single dose of daprodustat 4mg one tablet, administered orally in fasted state on Day 1 in intervention Period 2
Arm/Group | Daprodustat 4mg (Fed) | Daprodustat 4mg(Fasted)
Number analyzed (Participants) | 12 | 12
Hour*nanogram/milliliter
  AUC (0-t) | 142.9556 (18.0) | 156.4222 (19.3)
  AUC (0-inf) | 143.1156 (18.0) | 156.5481 (19.2)
Statistical Analysis 1: Comparison: Daprodustat 4mg (Fed) vs Daprodustat 4mg(Fasted); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric mean = 0.91, 90% CI 2-sided [0.82 to 1.01] — AUC (0-t)
Statistical Analysis 2: Comparison: Daprodustat 4mg (Fed) vs Daprodustat 4mg(Fasted); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric mean = 0.91, 90% CI 2-sided [0.82 to 1.01] — AUC (0-inf)

10. Primary Outcome: Part 2: Cmax of Daprodustat
Description: as for outcome 3
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12hours post-dose on Day 1, 24hours post-dose on Day 2
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter (ng/L)
Groups:
- Daprodustat 4mg Fed: Participants received a single dose of daprodustat 4mg one tablet, administered orally in fed state on Day 1 in intervention period 1
- Daprodustat 4mg Fasted: Participants received single dose of daprodustat 4mg one tablet, administered orally in fasted state on Day 1 in intervention Period 2
Arm/Group | Daprodustat 4mg Fed | Daprodustat 4mg Fasted
Number analyzed (Participants) | 12 | 12
Nanogram/milliliter (ng/L) | 67.8240 (26.7) | 76.1944 (29.8)
Statistical Analysis 1: Comparison: Daprodustat 4mg Fed vs Daprodustat 4mg Fasted; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geomtric mean = 0.89, 90% CI [0.73 to 1.08]

11. Primary Outcome: Part 2: T1/2 and MRT of Daprodustat
Description: Blood samples were collected at indicated time points and PK analysis was performed. PK parameters were determined by non-compartmental methods with Phoenix WinNonlin version 6.3.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12hours post-dose on Day 1, 24hours post-dose on Day 2
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Groups:
- Part 2: Daprodustat 4mg Fasted: Participants received single dose of daprodustat 4mg one tablet, administered orally in fasted state on Day 1 in intervention Period 2
Arm/Group | Daprodustat 4mg Fed | Part 2: Daprodustat 4mg Fasted
Number analyzed (Participants) | 12 | 12
hour
  t1/2 | 3.2160 (9.7) | 3.2389 (8.0)
  MRT | 3.2420 (25.2) | 2.6695 (26.8)

12. Primary Outcome: Part 2: Tmax of Daprodustat
Description: as for outcome 3
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12 hours post-dose on Day 1, 24 hours post-dose on Day 2
Population: PK Population.
Measure: Median (Full Range); unit: hour
Groups:
- Part 2: Daprodustat 4mg Fed: Participants received a single dose of daprodustat 4mg one tablet, administered orally in fed state on Day 1 in intervention period 1
Arm/Group | Part 2: Daprodustat 4mg Fed | Part 2: Daprodustat 4mg Fasted
Number analyzed (Participants) | 12 | 12
hour | 2.750 [1.00 to 3.00] | 1.750 [1.00 to 4.00]

13. Primary Outcome: Part 2: Percentage AUCex of Dapordustat
Description: as for outcome 3
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12 hours post-dose on Day 1, 24 hours post-dose on Day 2
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUCex
Groups:
- Part 2: Daprodustat 4mg Fed: Participants received a single dose of daprodustat 2mg*2 tablets, administered orally in fasted state on Day 1 in either of period 1 and Period 2 as per the randomization schedule
Arm/Group | Part 2: Daprodustat 4mg Fed | Part 2: Daprodustat 4mg Fasted
Number analyzed (Participants) | 12 | 12
Percentage of AUCex | 0.1071 (30.9) | 0.0723 (47.9)

14. Primary Outcome: Part 2: CL/F of Daprodustat
Description: as for outcome 3
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12 hours post-dose on Day 1, 24 hours post-dose on Day 2
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part 2: Daprodustat 4mg Fed | Part 2: Daprodustat 4mg Fasted
Number analyzed (Participants) | 12 | 12
Liters per hour | 27.9494 (18.0) | 25.5512 (19.2)

15. Primary Outcome: Part 2: Vz/F of Daprodustat
Description: as for outcome 3
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12 hours post-dose on Day 1, 24 hours post-dose on Day 2
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliters (mL)
Arm/Group | Part 2: Daprodustat 4mg Fed | Part 2: Daprodustat 4mg Fasted
Number analyzed (Participants) | 12 | 12
Milliliters (mL) | 129676.9 (18.7) | 119394.6 (19.7)

16. Primary Outcome: Part 2: Kel of Daprodustat
Description: as for outcome 3
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12 hours post-dose on Day 1, 24 hours post-dose on Day 2
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per hour
Arm/Group | Part 2: Daprodustat 4mg Fed | Part 2: Daprodustat 4mg Fasted
Number analyzed (Participants) | 12 | 12
Per hour | 0.2155 (9.7) | 0.2140 (8.0)

17. Secondary Outcome: Part 1: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant. Safety population comprised of all randomized participants who took at least one dose of study treatment.
Time Frame: Up to Day 16
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
Participants
  Any AE | 3 | 1
  Any SAE | 0 | 0

18. Secondary Outcome: Part 1: Change From Baseline Chemistry Paramters: Glucose, Calcium, Cholesterol, Chloride, High Density Lipoprotein (HDL) Cholesterol, Low Density Lipoprotein (LDL) Cholesterol, Potassium, Phosphate, Sodium, Triglycerides, and Urea.
Description: Blood samples were collected to analyze the chemistry parameters; glucose, calcium, cholesterol, chloride, HDL cholesterol, LDL cholesterol, potassium, phosphate, sodium, triglycerides, and urea. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the Post-Dose visit value.
Time Frame: Baseline (Day -1), 24hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimoles per Liter (mmol/L)
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
Millimoles per Liter (mmol/L)
  Glucose 24hours | -0.007619 (0.3094690) | -0.004270 (0.3243933)
  Calcium 24hours | -0.016144 (0.0694710) | -0.015834 (0.0623072)
  Cholesterol 24hours | -0.043607 (0.3197656) | 0.046747 (0.2952955)
  Chloride 24hours | 0.9 (1.74) | 0.5 (1.63)
  HDL cholesterol 24hours | -0.128793 (0.1230991) | -0.111397 (0.1067511)
  LDL cholesterol 24hours | 0.022818 (0.2151606) | 0.099462 (0.2265669)
  Potassium 24hours | 0.04 (0.295) | 0.03 (0.272)
  Phosphate 24hours | -0.102568 (0.1114273) | -0.091281 (0.1110710)
  Sodium 24hours | 0.2 (1.37) | 0.0 (1.50)
  Triglycerides 24hours | 0.21802 (0.273901) | 0.16385 (0.274955)
  Urea 24hours | -0.14000 (0.767902) | -0.29178 (0.840240)

19. Secondary Outcome: Part 1: Change From Baseline in Chemistry Parameters: Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Creatine Kinase, Lactate Dehydrogenase and Gamma Glutamyl Transferase (GGT).
Description: Blood samples were collected to analyze the chemistry parameters; ALP, ALT, AST, creatine kinase, lactate dehydrogenase and GGT. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the Post-Dose visit value.
Time Frame: Baseline (Day -1), 24hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: International unit per liter (IU/L)
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
International unit per liter (IU/L)
  ALP 24hours | -9.5 (17.24) | -10.8 (12.83)
  ALT 24hours | -2.0 (3.65) | -1.0 (3.19)
  AST 24hours | -2.1 (3.19) | -1.8 (3.22)
  Creatine kinase 24hours | -33.9 (28.73) | -32.3 (30.24)
  GGT 24hours | -1.6 (2.34) | -1.1 (1.34)
  Lactate dehydrogenase 24hours | -20.5 (12.30) | -19.2 (9.15)

20. Secondary Outcome: Part 1: Change From Baseline in Chemistry Parameters; Albumin, Protein.
Description: Blood samples were collected to analyze the chemistry parameters; albumin, protein. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the Post-Dose visit value.
Time Frame: Baseline (Day -1), 24hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
Grams per liter (g/L)
  Albumin 24hours | -2.0 (1.74) | -2.0 (1.69)
  Protein 24hours | -2.3 (2.90) | -2.1 (2.35)

21. Secondary Outcome: Part 1: Change From Baseline in Chemistry Parameters; Direct Bilirubin, Bilirubin, Creatinine, Urate
Description: Blood samples were collected to analyze the chemistry parameters; direct bilirubin, bilirubin, creatinine, urate. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the Post-Dose visit value.
Time Frame: Baseline (Day -1), 24hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
Micromoles per liter (umol/L)
  Direct bilirubin 24hours | 0.268 (0.7151) | 0.164 (0.6989)
  Bilirubin 24hours | 2.615 (5.0537) | 2.960 (4.7784)
  Creatinine 24hours | 1.7160 (4.18539) | 1.4110 (4.84901)
  Urate 24hours | 26.1245 (28.30344) | 25.6222 (28.35581)

22. Secondary Outcome: Part 1:Change From Baseline in Hematology Parameter; Hematocrit
Description: Blood samples were collected to analyze hematology parameters; hematocrit, reticulocytes. Platelets. Day-1 (one day before the Pre-Dose) was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the Post-Dose visit value.
Time Frame: Baseline (Day -1), 24hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
Proportion of red blood cells in blood | 0.0005 (0.01593) | 0.0014 (0.01464)

23. Secondary Outcome: Part 1:Change From Baseline in Hematology Parameter; Reticulocytes
Description: Blood samples were collected to analyze hematology parameters; reticulocytes. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the Post-Dose visit value.
Time Frame: Baseline (Day -1), 24hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Praportion of reticulocytes in blood
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
Praportion of reticulocytes in blood | -0.0005 (0.00179) | -0.0001 (0.00189)

24. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameters; Hemoglobin (Hb), Erythrocyte Mean Corpuscular Hb Concentration (MCHC)
Description: Blood samples were collected to analyze hematology parameters; Hb, EMCH concentration. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the Post-Dose visit value.
Time Frame: Baseline (Day -1), 24hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per Liter (g/L)
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
Grams per Liter (g/L)
  Hb 24hours | 1.1 (5.81) | 0.8 (4.99)
  MCHC 24hours | 2.1 (4.23) | 0.8 (4.99)

25. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameters; Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils
Description: Blood samples were collected to analyze hematology parameters; basophils, eosinophils, lymphocytes, monocytes, neutrophil. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the Post-Dose visit value.
Time Frame: Baseline (Day -1), 24hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Percentage of cells
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
Percentage of cells
  Basophils 24hours | -0.01 (0.173) | 0.00 (0.197)
  Eosinophils 24hours | 0.27 (0.871) | 0.25 (0.874)
  Lymphocytes 24hours | -1.47 (6.070) | -0.86 (7.049)
  Monocytes 24hours | -0.43 (1.293) | -0.33 (1.108)
  Neutrophils 24hours | 1.64 (6.407) | 0.94 (7.480)

26. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameter Erythrocyte MCHC
Description: Blood samples were collected to analyze hematology parameter; EMCH. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the Post-Dose visit value.
Time Frame: Baseline (Day -1), 24hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Picograms (pg)
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
Picograms (pg) | 0.11 (0.331) | 0.01 (0.319)

27. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameter Erythrocyte Mean Corpuscular Volume (EMCV)
Description: Blood samples were collected to analyze hematology parameter; EMCV. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the Post-Dose visit value.
Time Frame: Baseline (Day -1), 24hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
Femtoliters | -0.2 (0.75) | -0.2 (0.83)

28. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameters Platelets, Leukocytes
Description: Blood samples were collected to analyze hematology parameter; platelets, leukocytes. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the Post-Dose visit value.
Time Frame: Baseline (Day -1), 24hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Billion cells per liter (10^9/L)
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
Billion cells per liter (10^9/L)
  Platelets 24hours | 0.7 (13.21) | 2.0 (14.97)
  Leukocytes 24hours | -0.55 (0.883) | -0.53 (0.928)

29. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameter: Erythrocytes
Description: Blood samples were collected to analyze hematology parameter; erythrocytes. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the Post-Dose visit value.
Time Frame: Baseline (Day -1), 24hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Trillion cells/liter (10^12 cell/L)
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
Trillion cells/liter (10^12 cell/L) | 0.018 (0.1941) | 0.023 (0.1771)

30. Secondary Outcome: Part 1: Change From Baseline in Urinalysis Parameter; Potential of Hydrogen (pH)
Description: Urinary pH measurement is a routine part of urinalysis. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0). Urine samples were collected for the measurement of urine pH by method up to 24 hours in Part 1.Day-1 (one day before the Pre-Dose) was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the Post-Dose visit value.
Time Frame: Baseline (Day -1), 24hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
pH | -0.04 (0.573) | -0.07 (0.714)

31. Secondary Outcome: Part 1: Change From Baseline in Urinalysis Parameter; Specific Gravity
Description: Urinary specific gravity measurement is a routine part of urinalysis. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The concentration of the excreted molecules determines the urine's specific gravity. Urine samples were collected for the measurement of urine specific gravity by dipstick method up to 24 hours in Part 1. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the Post-Dose visit value.
Time Frame: Baseline (Day -1), 24hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Kilogram per cubic meter
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
Kilogram per cubic meter | 0.0092 (0.00744) | 0.0088 (0.00767)

32. Secondary Outcome: Part 1: Change From Baseline in Vital Signs; Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: DBP and SBP were measured in semi-supine position after 5 minutes rest for the participants at indicated time points. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -1), 3 and 24 hours (post-dose)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
Millimeters of mercury (mmHg)
  DBP 3hours | -2.9 (5.84) | -1.5 (7.00)
  DBP 24hours | -1.8 (6.38) | 0.1 (7.67)
  SBP 3hours | -0.6 (7.48) | -0.4 (7.92)
  SBP 24hours | -0.9 (8.07) | 0.2 (8.93)

33. Secondary Outcome: Part 1: Change From Baseline in Pulse Rate
Description: Pulse rate was measured in semi-supine position after 5 minutes rest for the participants at indicated time points. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -1), 3 and 24 hours (post-dose)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
Beats per minute
  Pulse rate 3hours | 0.0 (6.91) | 0.7 (4.78)
  Pulse rate 24hours | 0.1 (6.04) | 1.0 (5.12)

34. Secondary Outcome: Part 1: Change From Baseline in Temperature
Description: Temperature was measured in semi-supine position after 5 minutes rest for the participants at indicated time points. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -1), 3 and 24 hours (post-dose)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Celcius (c)
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
Celcius (c)
  Temperature 3hours | 0.23 (0.256) | 0.22 (0.311)
  Temperature 24hours | 0.10 (0.212) | 0.05 (0.330)

35. Secondary Outcome: Part 1: Change From Baseline in Electrocardiogram (ECG) Parameter; Mean Heart Rate (HR)
Description: Single 12-lead ECG's were obtained from using an ECG machine that automatically calculated the heart rate and measured PR Interval, QRS Duration, Uncorrected QT interval and Corrected QT (Fridericia's correction) interval at given time point. Day -1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -1), 3 and 24 hours (post-dose)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
Beats per minute
  Mean HR 3hours | 0.6 (5.01) | 0.2 (4.21)
  Mean HR 24hours | 1.2 (4.28) | 0.8 (5.18)

36. Secondary Outcome: Part 1: Change From Baseline in ECG Parameter; PR Interval, QRS Interval, QT Interval, QT Duration Corrected for Heart Rate by Friderician Formula (QTcF) Interval
Description: as for outcome 35
Time Frame: Baseline (Day -1), 3 and 24 hours (post-dose)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milliseconds (msec)
Arm/Group | Part 1: Daprodustat 2mg*2 | Part 1: Daprodustat 4mg*1
Number analyzed (Participants) | 51 | 52
Milliseconds (msec)
  PR Interval, Aggregate 3hours | -3.3 (10.87) | -3.8 (9.40)
  PR Interval, Aggregate 24hours | 1.4 (8.13) | 0.0 (12.55)
  QRS Duration, Aggregate 3hours | -2.8 (6.50) | -1.5 (6.42)
  QRS Duration, Aggregate 24hours | -1.6 (6.62) | 0.2 (6.50)
  QT interval, Aggregate 3hours | 0.0 (20.31) | 0.8 (17.63)
  QT interval, Aggregate 24hours | -5.2 (17.42) | -5.3 (18.33)
  QTcF interval, Aggregate 3hours | 1.2 (14.98) | 1.6 (14.73)
  QtcF Interval, Aggregate 24hours | -2.4 (13.65) | -3.1 (13.70)

37. Secondary Outcome: Part 2: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: as for outcome 17
Time Frame: Up to Day 16
Population: Safety Population
Measure: Number; unit: Participants
Groups:
- Part 2: Daprodustat 4mg (Fed): Participants received a single dose of daprodustat 4mg one tablet, administered orally in fed state on Day 1 in intervention period 1, the washout between the 2 intervention periods was set to be ≥ 5 days
- Part 2: Daprodustat 4mg (Fasted): Participants received single dose of Daprodustat 4mg one tablet, administered orally in fasted state on Day 1 in intervention Period 2
Arm/Group | Part 2: Daprodustat 4mg (Fed) | Part 2: Daprodustat 4mg (Fasted)
Number analyzed (Participants) | 12 | 12
Participants
  Any AE | 0 | 0
  Any SAE | 0 | 0

38. Secondary Outcome: Part 2: Change From Baseline Chemistry Parameters; Glucose, Calcium, Cholesterol, Chloride, HDL Cholesterol, LDL Cholesterol, Potassium, Phosphate, Sodium, Triglycerides, and Urea
Description: Blood samples were collected to analyze the chemistry parameters; glucose, calcium, cholesterol, chloride, HDL cholesterol, LDL cholesterol, potassium, phosphate,sodium, triglycerides, and urea. Day-1 (one day before the Pre-Dose) was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the Post-Dose visit value.
Time Frame: Baseline (Day -1), 24 hours (post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimoles per Liter (mmol/L)
Arm/Group | Part 2: Daprodustat 4mg (Fed) | Part 2: Daprodustat 4mg (Fasted)
Number analyzed (Participants) | 12 | 12
Millimoles per Liter (mmol/L)
  Glucose, 24hours | -0.425577 (0.2902134) | -0.018503 (0.2530908)
  Calcium, 24hours | -0.076929 (0.0515273) | -0.058217 (0.0595515)
  Cholesterol, 24hours | -0.172400 (0.2567913) | -0.094820 (0.2225472)
  Chloride, 24hours | 1.5 (1.45) | 2.1 (2.27)
  HDL cholesterol, 24hours | -0.165935 (0.0995210) | -0.148695 (0.0826086)
  LDL cholesterol, 24hours | -0.170245 (0.1823445) | -0.066805 (0.1724049)
  Potassium, 24hours | 0.06 (0.294) | 0.19 (0.231)
  Phosphate, 24hours | -0.029599 (0.0928311) | -0.080725 (0.1324212)
  Sodium, 24hours | 0.3 (2.35) | 0.9 (1.38)
  Triglycerides, 24hours | 0.25331 (0.219827) | 0.08475 (0.197228)
  Urea, 24hours | 0.19040 (0.552713) | -0.14875 (0.588353)

39. Secondary Outcome: Part 2: Change From Baseline in Chemistry Paremeters; ALP, ALT, AST, Creatine Kinase, Lactate Dehydrogenase, GGT
Description: Blood samples were collected to analyze the chemistry parameters; ALP,ALT, AST, creatine kinase, lactate dehydrogenase and GGT. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the Post-Dose visit value.
Time Frame: Baseline (Day -1), 24 hours (post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International unit per liter (IU/L)
Arm/Group | Part 2: Daprodustat 4mg (Fed) | Part 2: Daprodustat 4mg (Fasted)
Number analyzed (Participants) | 12 | 12
International unit per liter (IU/L)
  ALP, 24hours | -18.9 (15.48) | -13.3 (10.54)
  ALT, 24hours | -3.1 (2.43) | -3.5 (2.02)
  AST, 24hours | -2.8 (2.18) | -2.7 (2.46)
  Creatine kinase, 24hours | -28.3 (13.70) | -15.3 (17.56)
  Lactate dehydrogenase, 24hours | -21.0 (9.68) | -18.4 (9.05)
  GGT, 24hours | -1.0 (1.41) | -1.6 (2.11)

40. Secondary Outcome: Part 2: Change From Baseline in Chemistry Parameters; Albumin, Protein
Description: as for outcome 20
Time Frame: Baseline (Day -1), 24 hours (post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Part 2: Daprodustat 4mg (Fed) | Part 2: Daprodustat 4mg (Fasted)
Number analyzed (Participants) | 12 | 12
Grams per liter (g/L)
  Albumin 24hours | -3.2 (1.34) | -1.9 (1.16)
  Protein 24hours | -3.4 (2.94) | -2.6 (2.02)

41. Secondary Outcome: Part 2: Change From Baseline in Chemistry Parameters; Direct Bilirubin, Bilirubin, Creatinine, Urate
Description: as for outcome 21
Time Frame: Baseline (Day -1), 24 hours (post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | Part 2: Daprodustat 4mg (Fed) | Part 2: Daprodustat 4mg (Fasted)
Number analyzed (Participants) | 12 | 12
Micromoles per liter (umol/L)
  Direct bilirubin, 24hours | 0.000 (0.000) | 0.000 (1.0312)
  Bilirubin, 24hours | 2.280 (5.2748) | 1.425 (3.1643)
  Creatinine, 24hours | -1.6207 (5.16603) | -1.1050 (5.68072)
  Urate, 24hours | 23.2963 (20.98470) | 21.8093 (19.53615)

42. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameters; Hematocrit
Description: Blood samples were collected to analyze hematology parameter; hematocrit. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the Post-Dose visit value.
Time Frame: Baseline (Day -1), 24 hours (post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Praportion of red blood cells in blood
Arm/Group | Part 2: Daprodustat 4mg (Fed) | Part 2: Daprodustat 4mg (Fasted)
Number analyzed (Participants) | 12 | 12
Praportion of red blood cells in blood | -0.0052 (0.01629) | -0.0025 (0.01519)

43. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameters; Reticulocytes
Description: Blood samples were collected to analyze hematology parameter; reticulocytes. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the Post-Dose visit value.
Time Frame: Baseline (Day -1), 24 hours (post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Praportion of reticulocytes in blood
Arm/Group | Part 2: Daprodustat 4mg (Fed) | Part 2: Daprodustat 4mg (Fasted)
Number analyzed (Participants) | 12 | 12
Praportion of reticulocytes in blood | -0.0002 (0.00164) | -0.0010 (0.00186)

44. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameters; Hb, Erythrocyte MCHC
Description: Blood samples were collected to analyze hematology parameters; Hb, erythrocyte MCHC. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the Post-Dose visit value.
Time Frame: Baseline (Day -1), 24 hours (post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Part 2: Daprodustat 4mg (Fed) | Part 2: Daprodustat 4mg (Fasted)
Number analyzed (Participants) | 12 | 12
Grams per liter (g/L)
  Hb 24hours | -2.1 (5.28) | -1.2 (5.37)
  EMCH concentration 24hours | 0.4 (5.55) | -0.6 (4.66)

45. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameters; Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils
Description: Blood samples were collected to analyze hematology parameters; basophils, eosinophils, lymphocytes, monocytes, neutrophils. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the Post-Dose visit value.
Time Frame: Baseline (Day -1), 24 hours (post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percentage of cells
Arm/Group | Part 2: Daprodustat 4mg (Fed) | Part 2: Daprodustat 4mg (Fasted)
Number analyzed (Participants) | 12 | 12
Percentage of cells
  Basophils, 24hours | -0.04 (0.193) | -0.17 (0.239)
  Eosinophils, 24hours | 0.62 (1.620) | -0.49 (0.312)
  Lymphocytes, 24hours | -2.31 (3.815) | -1.14 (6.015)
  Monocytes, 24hours | -0.38 (0.732) | -0.03 (1.414)
  Neutrophils, 24hours | 2.12 (5.072) | 1.83 (5.829)

46. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: EMCH
Description: as for outcome 26
Time Frame: Baseline (Day -1), 24 hours (post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: picograms
Arm/Group | Part 2: Daprodustat 4mg (Fed) | Part 2: Daprodustat 4mg (Fasted)
Number analyzed (Participants) | 12 | 12
picograms | 0.10 (0.413) | 0.03 (0.311)

47. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter EMCV
Description: as for outcome 27
Time Frame: Baseline (Day -1), 24 hours (post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Part 2: Daprodustat 4mg (Fed) | Part 2: Daprodustat 4mg (Fasted)
Number analyzed (Participants) | 12 | 12
Femtoliters | 0.5 (0.67) | 0.3 (0.97)

48. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameters Platelets, Leukocytes
Description: as for outcome 28
Time Frame: Baseline (Day -1), 24 hours (post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Billion cells per liter (10^9/L)
Arm/Group | Part 2: Daprodustat 4mg (Fed) | Part 2: Daprodustat 4mg (Fasted)
Number analyzed (Participants) | 12 | 12
Billion cells per liter (10^9/L)
  Platelets, 24hours | -10.9 (11.19) | -3.2 (12.04)
  Leukocytes, 24hours | -0.27 (0.780) | -0.39 (0.579)

49. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter Erythrocytes
Description: as for outcome 29
Time Frame: Baseline (Day -1), 24 hours (post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Trillion cells/liter (10^12 cell/L)
Arm/Group | Part 2: Daprodustat 4mg (Fed) | Part 2: Daprodustat 4mg (Fasted)
Number analyzed (Participants) | 12 | 12
Trillion cells/liter (10^12 cell/L) | -0.083 (0.1859) | -0.044 (0.1767)

50. Secondary Outcome: Part 2: Change From Baseline in Urinalysis Parameter; Potential of Hydrogen (pH)
Description: Urinary pH measurement is a routine part of urinalysis. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0). Urine samples were collected for the measurement of urine pH by method up to 24 hours in Part 2. Day-1 (one day before the Pre-Dose) was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the Post-Dose visit value.
Time Frame: Baseline (Day -1), 24 hours (post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 2: Daprodustat 4mg (Fed) | Part 2: Daprodustat 4mg (Fasted)
Number analyzed (Participants) | 12 | 12
pH | 0.13 (0.433) | 0.13 (0.608)

51. Secondary Outcome: Part 2: Change From Baseline in Urinalysis Parameter; Specific Gravity
Description: Urinary specific gravity measurement is a routine part of urinalysis. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The concentration of the excreted molecules determines the urine's specific gravity. Urine samples were collected for the measurement of urine specific gravity by dipstick method up to 24 hours in Part 2. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the Post-Dose visit value.
Time Frame: Baseline (Day -1), 24 hours (post-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Kilogram per cubic meter
Arm/Group | Part 2: Daprodustat 4mg (Fed) | Part 2: Daprodustat 4mg (Fasted)
Number analyzed (Participants) | 12 | 12
Kilogram per cubic meter | 0.0054 (0.01215) | 0.0013 (0.00900)

52. Secondary Outcome: Part 2: Change From Baseline in Vital Signs; Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: DBP and SBP were measured in semi-supine position after 5 minutes rest for the participants at indicated time point. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -1),3 and 24hours (pre-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Part 2: Daprodustat 4mg (Fed) | Part 2: Daprodustat 4mg (Fasted)
Number analyzed (Participants) | 12 | 12
Millimeters of mercury (mmHg)
  DBP, 3hours | -4.8 (4.90) | 0.2 (5.61)
  DBP, 24hours | -0.6 (7.14) | 2.8 (6.97)
  SBP, 3hours | 0.7 (6.10) | -1.3 (8.41)
  SBP, 24hours | 1.4 (6.93) | 1.3 (5.18)

53. Secondary Outcome: Part 2: Change From Baseline in Pulse Rate
Description: Pulse rate was measured in semi-supine position after 5 minutes rest for the participants at indicated time points. Day -1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -1),3 and 24hours (pre-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 2: Daprodustat 4mg (Fed) | Part 2: Daprodustat 4mg (Fasted)
Number analyzed (Participants) | 12 | 12
Beats per minute
  Pulse rate, 3hours | 6.1 (5.37) | -1.5 (5.82)
  Pulse rate, 24hours | 4.0 (5.24) | 2.9 (6.05)

54. Secondary Outcome: Part 2: Change From Baseline in Temperature
Description: Temperature was measured in semi-supine position after 5 minutes rest for the participants at indicated time points. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day -1),3 and 24hours (pre-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: celcius
Arm/Group | Part 2: Daprodustat 4mg (Fed) | Part 2: Daprodustat 4mg (Fasted)
Number analyzed (Participants) | 12 | 12
celcius
  Temperature, 3hours | 0.28 (0.302) | 0.13 (0.293)
  Temperature, 24hours | 0.02 (0.424) | 0.03 (0.245)

55. Secondary Outcome: Part 2: Change From Baseline in ECG Parameter; Mean Heart Rate (HR)
Description: as for outcome 35
Time Frame: Baseline (Day -1),3 and 24hours (pre-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Part 2: Daprodustat 4mg (Fed) | Part 2: Daprodustat 4mg (Fasted)
Number analyzed (Participants) | 12 | 12
Beats/minute
  Mean HR, 3hours | 3.7 (6.18) | 0.0 (4.07)
  Mean HR, 24hours | 3.1 (6.60) | 0.6 (4.72)

56. Secondary Outcome: Part 2: Change From Baseline in ECG Parameter; PR Interval, QRS Interval, QT Interval, QTcF Interval
Description: as for outcome 35
Time Frame: Baseline (Day -1),3 and 24hours (pre-dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milliseconds (msec)
Arm/Group | Part 2: Daprodustat 4mg (Fed) | Part 2: Daprodustat 4mg (Fasted)
Number analyzed (Participants) | 12 | 12
Milliseconds (msec)
  PR Interval, Aggregate, 3hours | -6.2 (6.00) | -2.7 (9.55)
  PR Interval, Aggregate, 24hours | -4.0 (7.53) | -3.2 (7.11)
  QRS Duration, Aggregate, 3hours | -1.5 (4.52) | -0.5 (5.13)
  QRS Duration, Aggregate, 24hours | -0.8 (4.39) | 2.8 (7.93)
  QT interval, Aggregate, 3hours | -13.0 (15.81) | 1.0 (16.28)
  QT Interval, Aggregate, 24hours | -7.3 (13.73) | -2.2 (12.34)
  QTcF Interval, Aggregate, 3hours | -5.3 (11.93) | 1.2 (13.64)
  QTcF Interval, Aggregate, 24hours | -0.6 (12.87) | -1.1 (9.69)

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the Day -1 up to follow-up ( 16 days for Part 1 and Part 2)
Description: Safety Population was used. Safety Population comprised of all participants who received at least one dose of a study treatment.
Groups:
- Daprodustat 2mg*2 Followed by Daprodustat 4mg*1: Participants received a single dose Daprodustat 2 milligram (mg) two tablets followed by Daprodustat 4 mg single tablet, administered orally on Day 1.
- Daprodustat 4mg*1 Tablet Followed by Daprodustat 2mg*2tablets: Participants received a single dose Daprodustat 4 mg one tablet followed by Daprodustat 2 mg two tablets, administered orally on Day 1.
- Daprodustat 4mg*1 (Fed) Followed by Daprodustat 4mg*1 (Fasted): Participants received a single dose Daprodustat 4 mg one tablet in fed state followed by Daprodustat 4 mg one tablet as single dose in fasted state, administered orally on Day 1.
- Daprodustat 4mg*1 (Fasted) Followed by Daprodustat 4mg*1(Fed): Participants received a single dose Daprodustat 4 mg one tablet in fasted state followed by Daprodustat 4 mg one tablet as single dose in fed state, administered orally on Day 1.
Arm/Group | Daprodustat 2mg*2 Followed by Daprodustat 4mg*1 | Daprodustat 4mg*1 Tablet Followed by Daprodustat 2mg*2tablets | Daprodustat 4mg*1 (Fed) Followed by Daprodustat 4mg*1 (Fasted) | Daprodustat 4mg*1 (Fasted) Followed by Daprodustat 4mg*1(Fed)
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/52 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/52 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/51 | 1/52 | 0/12 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daprodustat 2mg*2 Followed by Daprodustat 4mg*1 (N=51) | Daprodustat 4mg*1 Tablet Followed by Daprodustat 2mg*2tablets (N=52) | Daprodustat 4mg*1 (Fed) Followed by Daprodustat 4mg*1 (Fasted) (N=12) | Daprodustat 4mg*1 (Fasted) Followed by Daprodustat 4mg*1(Fed) (N=12)
Tonsilitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT03493386/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/86/NCT03493386/SAP_001.pdf